CLINICAL TRIAL: NCT07405203
Title: A Single-Arm Pilot Study to Assess Safety and Performance of the EndoR Surgical System to Perform Endoscopic Submucosal Dissection (ESD) for the Treatment of Colorectal Lesions
Brief Title: Assessment of the EndoR System in ESD for Colorectal Lesions
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Hon Chi Yip, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRE-2025.546
Record Dates: First submitted 2026-02-04; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Colorectal Lesions
Keywords: EndoR; ESD; Endoscopic Submucosal Dissection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EndoR System assisted ESD (Experimental): Recruited subjects will undergo robotic ESD under general anesthesia using EndoR Surgical System.
  Interventions: Device: EndoR Surgical System

INTERVENTIONS:
Device: EndoR Surgical System — The EndoR Surgical System is a master-slave robotic platform designed for endoscopic surgery, featuring flexible dual arms and cognitive control system.

SUMMARY:
Gastrointestinal (GI) cancers are common and significant causes of cancer death worldwide. GI cancers grow from the mucosal layer. If pre-malignant and early cancers are removed en bloc at an early stage before they spread to lymph nodes, survival rates can be improved.

Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) were developed as minimally invasive, organ-sparing methods for removing pre-malignant and early GI cancers. While EMR is suitable for smaller lesions, ESD is typically required for larger lesions. ESD offers the advantage of a higher rate of complete, single-piece resection, which is associated with a lower risk of local recurrence compared to EMR. However, ESD is a technically complex procedure with a higher risk of complications, such as perforation and bleeding.

Conventional ESD is performed using a flexible endoscope with a single instrument channel to access the GI tract. This setup presents several challenges, including difficulty in maintaining the endoscope in a stable position, limited ability to provide effective tissue traction, and frequent intraprocedural bleeding. As a result, ESD demands a high level of technical skills from surgeons.

The EndoR Surgical System was developed to address these challenges, aiming to allow surgeons to operate two surgical instruments with enhanced dexterity and a broader range of motions. Both pre-clinical ex-vivo studies and in-vivo studies were conducted in the development of this surgical system.

Six pre-clinical ex-vivo studies were conducted in porcine stomach between 2015 and 2023 and eleven pre-clinical in-vivo studies were conducted in live porcine models with the lesion sites at stomach, rectum and left colon between 2016 and 2024. These pre-clinical studies were conducted in LASEC-PWH, MISSC-PWH and Hybrid Operating Room of Multi-Scale Medical Robotics Center (MRC) accordingly.

Based on data from the ex-vivo and in-vivo experiments, two key conclusions can be drawn:

i) After several training sessions, the operator's performance became more consistent and efficient.

ii) The dissection rate increased as the dissection area grew-a phenomenon not observed in conventional procedures using a single endoscope and dissection tool.

From the results demonstrated from the pre-clinical studies, the EndoR Surgical System allows for greater dexterity and precision in manipulating instruments, which is particularly advantageous for larger lesions. This precision can lead to more effective dissection and reduced damage to surrounding tissues. This may also reduce the risk of complications associated with ESD. By minimizing trauma to adjacent structures, the likelihood of adverse events, such as bleeding or perforation, may be significantly lowered. Patients may experience faster recovery times, contributing to improved patients' satisfaction and outcomes. As the risk of complications decreases, endoscopic procedures like ESD could become accessible to a broader patient population.

While performing ESD is generally considered safe, it still remains a technically demanding procedure with the assistance of the surgical robotic system. The use of surgical robots introduces the risk of equipment malfunctions, which can lead to complications during the procedure. Additionally, any technical issues may result in delays, potentially compromising patient safety.

The attending physicians will monitor and examine the subjects as necessary and appropriate and work carefully to ensure their safety. In the event of an adverse reaction, countermeasures will be taken as appropriate, and focus will be placed on ensuring the safety of the subjects while the cause of the reaction is investigated.

The objective of this study is to assess the safety and performance of the EndoR Surgical System for the treatment of patients with colorectal malignant lesions. Technical success, clinical success and any adverse events shall be recorded.

DETAILED DESCRIPTION:
Background Information

1. Purpose of the System 1.1. Device Name The EndoR Surgical System is a master-slave robotic platform designed for endoscopic surgery, featuring flexible dual arms and a cognitive control system.

   1.2. Intended Indications and Usage The EndoR Surgical System is an advanced endoscopic surgical robotic system designed to assist surgeons and endoscopists to perform endoscopic surgeries. This is a system intended to provide both visualization and therapeutic access to the adult gastrointestinal (GI) tract for endoscopic surgeries, aiming to improve visualization and potentially reduce procedure time and technical complexity.

   Comprehensive guidelines for the preparation and operation of the EndoR Surgical System are provided in the Instructions for Use (IFU). The IFU will be distributed to all investigators and reviewed during training prior to initiating any procedures.

   1.3. Product Description The EndoR Surgical System consists of two parts: the patient side and the surgeon side as shown in Figure 1. On the patient side, four main components can be found: a processing unit, a robotic carrier, a driving unit, and an overtube system with instruments. On the surgeon side, three main components can be found: a master console, a surgical monitor, and an ergonomic surgeon chair.

   On the surgeon side, the master console is the surgeon's primary interface with the EndoR Surgical System. It features intuitive controls that allow the surgeon to manipulate the robotic instruments with high precision remotely. The console transmits real-time commands to the patient-side processing unit. The surgical monitor displays high-definition, real-time video feeds from the endoscopic camera and other imaging sources. It provides the surgeon with a clear and detailed view of the operative field, enabling accurate navigation and decision-making throughout the procedure. The ergonomic surgeon chair is designed to maximize operator comfort and minimize fatigue during lengthy procedures. It features adjustable support for posture and armrests for stability while operating the console. A foot pedal of the electrocautery machine is usually placed near the surgeon's chair to control the electrocautery action of the dissector manipulator.

   On the patient side, the processing unit serves as the central "brain" of the system. It receives commands from the surgeon's console, interprets input signals, and coordinates the actions of all robotic components. This unit integrates real-time data processing, safety algorithms, and system diagnostics to ensure precise and synchronized movements during surgery. The robotic carrier is a stable platform designed to securely position and support the endoscopic instruments at the patient's bedside. It provides the structural framework for mounting the driving unit and endoscopic overtube system and can be adjusted for optimal alignment with the patient's anatomy. The carrier provides three standard motions to enable fine adjustment of the orientation of the instrument: translation along the overtube axial axis, rotational motion along the overtube axial axis, and up-down and left-right motion. The driving unit contains the actuators and motors that physically control the motion of the instruments. It translates digital commands from the processing unit into mechanical actions, such as rotation, insertion, or articulation of the endoscopic tools. The flexible endoscopic overtube system is designed to guide and protect the endoscope and instruments as they are advanced into the patient's gastrointestinal tract. Integrated within the overtube are instruments capable of performing complex surgical tasks such as tissue dissection and retraction. The endoscopic overtube system enhances stability and precision during endoscopic procedures.

   The connection between the overtube and the driving unit incorporates two attachment mechanisms. The first is a rotary attachment mechanism, which allows the overtube to be connected axially, enabling the orientation to be selected prior to installing the instruments. This design addresses surgical scenarios where the treatment area is extensive and, with conventional endoscopes, would typically require repositioning the patient during the procedure. Instead, the rotary mechanism permits the overtube to rotate and lock securely at four distinct angles, optimizing the surgical posture of the manipulator without the need to move the patient. This feature streamlines the workflow and shortens overall procedure time by eliminating unnecessary setup steps. The second is a sliding attachment mechanism, which allows the overtube to be connected from the side of the driving unit. This mechanism is not used in normal operating procedures but is used only in emergency situations, for example when the overtube needs to be removed instantly from the patient.

   The active bending section of the endoscopic overtube is controlled by knots. Two bending directions are provided (pitch and yaw direction), and the bending angles of each direction can be locked by pulling the knot in the direction out of the driving unit. The endoscopic channel enables the use of an endoscopic camera within the system, offering a clear view of the surgical location. The decoupled motion between the camera and the instruments further enhances the field of view and visual stability.
2. Findings From Pre-clinical Studies 2.1. Background of the Disease and Endoscopic Procedures Gastrointestinal cancers are common and significant causes of cancer death worldwide. GI cancers grow from the mucosal layer. If pre-malignant and early cancers are removed en bloc at an early stage before they spread to lymph nodes, survival rates can be improved.

   Endoscopic mucosal resection (EMR) and endoscopic submucosal dissection (ESD) were developed as minimally invasive, organ-sparing methods for removing pre-malignant and early gastrointestinal cancers. While EMR is suitable for smaller lesions, ESD is typically required for larger lesions. ESD offers the advantage of a higher rate of complete, single-piece resection, which is associated with a lower risk of local recurrence compared to EMR. However, ESD is a technically complex procedure with a higher risk of complications such as perforation and bleeding.

   Conventional ESD is performed using a flexible endoscope with a single instrument channel to access the gastrointestinal tract. This setup presents several challenges, including difficulty in maintaining the endoscope in a stable position, limited ability to provide effective tissue traction, and frequent intraprocedural bleeding. As a result, ESD demands a high level of technical skill from surgeons.

   2.2. Summary of Pre-clinical Studies The EndoR Surgical System was developed to address these challenges, aiming to allow surgeons to operate two surgical instruments with enhanced dexterity and a broader range of motions. Both pre-clinical ex-vivo studies and in-vivo studies were conducted in the development of this surgical system.

   Six pre-clinical ex-vivo studies were conducted in porcine stomach between 2015 and 2023, and eleven pre-clinical in-vivo studies were conducted in live porcine models with the lesion sites at the stomach, rectum, and left colon between 2016 and 2024. These pre-clinical studies were conducted in LASEC-PWH, MISSC-PWH, and the Hybrid Operating Room of the Multi-Scale Medical Robotics Center (MRC).

   I. Pre-clinical (Ex-vivo) Study Six pre-clinical ex-vivo studies were conducted between 2015 and 2023, spanning from the initial development of the robotic arms to the fully functional robotic platform. All studies utilized porcine stomach specimens in a bench-top setup.

   II. Pre-clinical (In-vivo) Study Eleven pre-clinical in-vivo studies were conducted between 2016 and 2024. All studies were performed in live porcine models weighing between 30 and 55 kg. The surgical sites included the stomach, rectum, and left colon. All studies were conducted under the supervision of clinical experts and were administered in a registered pre-clinical laboratory. The porcine models were given analgesics for pain relief before procedures and were euthanized before the end of the study if they suffered any serious injury or showed signs of severe pain or distress. Oxygen saturation and heart rate were monitored throughout the studies, and the porcine models were sacrificed by overdose of anesthetic.

   Based on data from the ex-vivo and in-vivo experiments, two key conclusions can be drawn:

   i) After several training sessions, operator performance became more consistent and efficient.

   ii) The dissection rate increased as the dissection area grew, a phenomenon not observed in conventional procedures using a single endoscope and dissection tool.
3. Potential Risks and Benefits From the results demonstrated in the pre-clinical studies, the EndoR Surgical System allows for greater dexterity and precision in manipulating instruments, which is particularly advantageous for larger lesions. This precision can lead to more effective dissection and reduced damage to surrounding tissues. This may also reduce the risk of complications associated with ESD. By minimizing trauma to adjacent structures, the likelihood of adverse events such as bleeding or perforation may be significantly lowered. Patients may experience faster recovery times, contributing to improved satisfaction and outcomes. As the risk of complications decreases, endoscopic procedures like ESD could become accessible to a broader patient population.

   While performing ESD is generally considered safe, it remains a technically demanding procedure even with the assistance of the surgical robotic system. The use of surgical robots introduces the risk of equipment malfunctions, which can lead to complications during the procedure. Additionally, any technical issues may result in delays, potentially compromising patient safety.

   The attending physicians will monitor and examine subjects as necessary and will work carefully to ensure subject safety. In the event of an adverse reaction, countermeasures will be taken as appropriate, and focus will be placed on ensuring subject safety while the cause of the reaction is investigated.
4. Duration of the Study and Follow-up Period The total duration of this study is two years. The enrollment period is expected to be completed within approximately one year, involving six subjects. Upon discharge, follow-up visits of subjects for this study will take place at the fourth to sixth week, sixth to eighth month, and twelfth to fourteenth month as clinically indicated. All subjects enrolled in this study will also receive clinical follow-up and surveillance according to standard clinical protocols thereafter.
5. Compliance

   This study will be conducted in compliance with the following guidelines and regulations:
   * International Council for Harmonization (ICH) Guideline on Good Clinical Practice (ICH E6)
   * Declaration of Helsinki
   * ISO 14155:2011 - Clinical Investigation of Medical Devices for Human Subjects (Good Clinical Practice)
   * All applicable local legal and regulatory requirements, as appropriate
6. Study Population This study will recruit six adult patients with superficial colorectal lesions scheduled for endoscopic submucosal dissection (ESD).

Trial Objective and Purpose

1. Objective The objective of this study is to assess the safety and performance of the EndoR Surgical System for the treatment of patients with colorectal malignant lesions. Technical success, clinical success, and any adverse events will be recorded.
2. Purpose The purpose of this study is to evaluate the EndoR Surgical System in human subjects. The EndoR Surgical System is designed for endoscopic procedures in the gastrointestinal (GI) tract through the natural orifices of the human body, with the goal of establishing a reliable, minimally invasive system that enhances patient outcomes.
3. Hypothesis The EndoR Surgical System is safe and efficacious for use in colonic endoscopic submucosal dissection.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 85.
* Patient with superficial colorectal lesions, scheduled for endoscopic submucosal dissection (ESD). According to the European Society of Gastrointestinal Endoscopy (ESGE) and the Japan Gastroenterological

Endoscopy Society (JGES) guidelines for colorectal ESD:

i. Lesions for which en bloc resection with snare EMR would be difficult to apply; ii. Mucosal tumors with submucosal fibrosis; iii. Sporadic tumors in conditions of chronic inflammation; iv. Local residual or recurrent early carcinomas after endoscopic resection.

Exclusion Criteria:

* No informed consent available.
* Carcinoma of colon or rectum with invasion to submucosa or beyond.
* Evidence of distant metastasis.
* Another active malignancy present.
* Pregnant.
* Patients are unfit for general anesthesia.
* The target lesion that could not be reached by the endoscopic platform.
* Have been recruited in another clinical trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-01-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of complete (R0) resection | 1 day
  Defined as en bloc, one-piece resection with histologically confirmed tumor-free lateral and vertical margins.
  Unit of measure: % of procedures

SECONDARY OUTCOMES:
[Safety] Rate of intraoperative bleeding | 1 day
  Bleeding at resection site prolonging procedure but not requiring transfusion or surgical intervention.
  Unit of measure: % of procedures
[Safety] Rate of adjunctive procedures | 1 day
  Rate of adjunctive procedures, during study procedure required to control bleeding (e.g. clips or haemostatic agents).
  Unit of measure: % of procedures
[Safety] All-cause mortality | 12 months
  Death from any cause within 12 months following the index procedure. Unit of measure: % of patients
[Safety] Rate of infection | 30 days
  Clinical sepsis with changes in inflammatory markers, as adjudicated by investigators.
  Unit of measure: % of patients
[Safety] Rate of Serious Adverse Events (SAEs) | 12 months
  Proportion of subjects experiencing any SAE during the index procedure, at discharge, or within 12 months.
  Unit of measure: % of patients
[Safety] Rate of SAEs - death | 12 months
  Death occurring within 12 months of index procedure. Unit of measure: % of patients
[Safety] Rate of SAEs - serious deterioration in the health | 12 months
  Rate of serious deterioration in the health of the subject, users, or other persons as defined by one or more of the following:
  i. a life-threatening illness or injury, or ii. a permanent impairment of a body structure or a body function including chronic diseases, or iii. in-patient or prolonged hospitalization, or iv. medical or surgical intervention to prevent life-threatening illness or injury, or permanent impairment to a body structure or a body function.
  Unit of measure: % of patients
[Safety] Rate of SAEs - fetal complications | 12 months
  Proportion of subjects experiencing fetal distress, fetal death, congenital abnormality, or birth defect (including physical or mental impairment) following the index procedure.
  Unit of measure: % of cases involving pregnancy
[Performance] Technical success rate | 30 days
  En bloc, one-piece excision of the neoplasm irrespective of histopathology, without device-related SAE through 30 days.
  Unit of measure: % of procedures
[Performance] Duration of instrument calibration | 1 day
  Total time for calibration of the device (e.g., dissector/retractor). Unit of measure: minutes
[Performance] Duration of resection | 1 day
  Time taken to complete neoplasm excision. Unit of measure: minutes
[Performance] Total ESD procedure time | 1 day
  Time from start of submucosal injection to end of procedure. Unit of measure: minutes
[Performance] Dissection rate | 1 day
  Rate at which the target tissue is dissected during ESD. Dissection rate = Resected lesion area / Dissection time Unit of measure: mm²/minute
[Performance] Histological analysis of resected specimen | 30 days
  Pathological evaluation of resected specimen for completeness, margin status, and depth of invasion.
  Unit of measure: categorical
[Performance] Proportion of time the submucosa was visualized | 1 day
  Proportion of time submucosa visualized during procedure (SM ratio) Unit of measure: % of total procedure time
[Performance] Number of additional submucosal injections required | 1 day
  Count of reinforcement injections used during procedure. Unit of measure: number per procedure
[Performance] Length of hospital stay | up to discharge
  Number of days from procedure to discharge. Unit of measure: days
[Performance] Rate of device deficiencies | 1 day
  Proportion of procedures affected by any device malfunction or use error. Unit of measure: % of procedures
[Performance] NASA Task Load Index | 1 day
  NASA Task Load Index (NASA-TLX) score reflecting perceived workload during the procedure (range 0-100; higher = greater workload).
  Unit of measure: score (0-100)
[Performance] Overall rate of intraprocedural adverse events | 1 day
  Rate of all intra-procedural adverse event. Unit of measure: % of procedures
[Performance] Rate of intraprocedural adverse events - partial thickness muscle damage | 1 day
  Partial-thickness muscle injury during procedure. Unit of measure: % of procedures
[Performance] Rate of intraprocedural adverse events - full thickness perforation | 1 day
  Full-thickness perforation during procedure. Unit of measure: % of procedures
[Performance] Rate of intraprocedural adverse events - hemorrhage | 1 day
  Major bleeding during the procedure requiring transfusion or causing >2 g/dL hemoglobin drop.
  Unit of measure: % of procedures
[Performance] Rate of intraprocedural adverse events - peritonitis | 1 day
  Inflammation of the peritoneum occurring intra-procedure. Unit of measure: % of procedures
[Performance] Rate of other intra-procedural adverse events | 1 day
  Any other intra-procedure adverse events not categorized above. Unit of measure: % of procedures
[Performance] Overall rate of postprocedural adverse events | 30 days
  Rate of all adverse events occurring after procedure. Unit of measure: % of patients
[Performance] Rate of postprocedural adverse events - electrocoagulation syndrome | 30 days
  Abdominal pain with fever or leukocytosis following procedure. Unit of measure: % of patients
[Performance] Rate of postprocedural adverse events - postoperative delayed bleeding | 30 days
  Bleeding after discharge requiring transfusion, intervention, or hemodynamic support.
  Unit of measure: % of patients
[Performance] Rate of postprocedural adverse events - post-procedure delayed perforation | 30 days
  Perforation occurring after completion of the index procedure. Unit of measure: % of patients
[Performance] Rate of other post-procedural adverse events | 30 days
  Any other adverse events related to the endoscopic procedure. Unit of measure: % of patients
[Performance] Colonoscopy findings at 6-8 months | 6-8 months post-procedure
  Colonoscopic analysis at the 6-8th month postoperative to assess:
  1. Healing of operative site
  2. Presence of suspicious tissue for biopsy (with results of biopsy)
  3. Presence of a stricture Unit of measure: categorical (healed / abnormal / stricture)
[Performance] Colonoscopy findings at 12-14 months | 12-14 months post-procedure
  Colonoscopic analysis at the 12-14th month postoperative to assess:
  1. Healing of operative site
  2. Presence of suspicious tissue for biopsy (with results of biopsy)
  3. Presence of a stricture Unit of measure: categorical (healed / abnormal / stricture)

OTHER OUTCOMES:
Rate of Major Adverse Events (MAE) | 30 days
  Composite safety endpoint defined as any of the following events within 30 days of the index procedure: bleeding requiring transfusion, discontinuation of the procedure, or open surgical control of hemorrhage; or perforation requiring endoscopic or surgical repair.
  Unit of measure: % of patients
Rate of intra-procedural bleeding (MAE) | 1 day
  Bleeding during the index procedure that requires transfusion, procedure discontinuation, or surgical intervention.
  Unit of measure: % of procedures
Rate of post-procedure perforation (MAE) | 30 days
  Perforation identified postoperatively and requiring endoscopic or surgical management.
  Unit of measure: % of patients
Rate of intra-procedural perforation (MAE) | 1 day
  Perforation recognized during the index procedure requiring adjunctive repair. Unit of measure: % of procedures
Rate of post-procedure bleeding (MAE) | 30 days
  Bleeding that occurs after the subject leaves the procedure room, requiring transfusion or surgical control.
  Unit of measure: % of patients

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Surgery, Faculty of Medicine, the Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akahoshi K, Akahane H, Murata A, Akiba H, Oya M. Endoscopic submucosal dissection using a novel grasping type scissors forceps. Endoscopy. 2007 Dec;39(12):1103-5. doi: 10.1055/s-2007-966842. PMID 18072064
- [Background] Teoh AY, Chiu PW, Wong SK, Sung JJ, Lau JY, Ng EK. Difficulties and outcomes in starting endoscopic submucosal dissection. Surg Endosc. 2010 May;24(5):1049-54. doi: 10.1007/s00464-009-0724-8. Epub 2009 Nov 13. PMID 19911227
- [Background] Oka S, Tanaka S, Kaneko I, Mouri R, Hirata M, Kawamura T, Yoshihara M, Chayama K. Advantage of endoscopic submucosal dissection compared with EMR for early gastric cancer. Gastrointest Endosc. 2006 Dec;64(6):877-83. doi: 10.1016/j.gie.2006.03.932. Epub 2006 Sep 20. PMID 17140890
- [Background] ASGE TECHNOLOGY COMMITTEE; Kantsevoy SV, Adler DG, Conway JD, Diehl DL, Farraye FA, Kwon R, Mamula P, Rodriguez S, Shah RJ, Wong Kee Song LM, Tierney WM. Endoscopic mucosal resection and endoscopic submucosal dissection. Gastrointest Endosc. 2008 Jul;68(1):11-8. doi: 10.1016/j.gie.2008.01.037. No abstract available. PMID 18577472
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842